CLINICAL TRIAL: NCT04345640
Title: The Spectrum and Profile of COVID-19 Infection and Its Impact on Liver - The Pan Asia-Pacific Prospective Multi-centre Observational Study (APCOLIS STUDY)
Brief Title: The Spectrum and Profile of COVID-19 Infection and Its Impact on Liver.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-COVID-01
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-04

CONDITIONS: Liver Cirrhoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid-19 with liver disease: Covid-19 with liver disease
  Interventions: Other: no intervention
- Covid-19 without liver disease: Covid-19 without liver disease
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
To address the existing deficiencies in the knowledge regarding liver involvement and spectrum of clinical presentation and the impact of COVID-19 infection in patients of liver disease was planned. The present study will be a hospital based and the cases of confirmed COVID-19 infection will be evaluated in relation to liver involvement irrespective of pre-existing liver disease. The primary objective was to address the clinical presentation, biochemical alteration and outcomes of COVID-19 infection in subjects with chronic hepatitis, cirrhosis in comparison to those having infection in the absence of pre-existing liver disease

ELIGIBILITY:
Inclusion Criteria:

1. All patients of COVID-19 positive
2. Age 18-70 years

Exclusion Criteria:

1. No Valid consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Covid-19 patients with or without liver disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Spontaneous recovery or death in both groups | 90 days

SECONDARY OUTCOMES:
Severity of prior as well as present decompensation in both groups | 90 days
Duration of prior as well as present decompensation in both groups | 90 days
Improvement in severity assessment Indices Model for End Stage Liver Disease (MELD) scores in both groups | 90 days
Improvement in severity assessment Indices Child-Turcotte-Pugh (CTP) scores in both groups | 90 days
Improvement in severity assessment Indices Sequential Organ Failure Assessment (SOFA) scores in both groups | 90 days
Improvement in severity assessment Indices Acute Physiology And Chronic Health Evaluation (APACHE) scores II in both groups | 90 days
Improvement in severity assessment Indices Chronic Liver Failure-Sequential Organ Failure Assessment (CLIF SOFA) scores in both groups. | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided